CLINICAL TRIAL: NCT05757128
Title: Optimizing Mental Health for Young People at Clinical High Risk for Psychosis (CHR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 063/2022
Record Dates: First submitted 2023-01-26; First posted 2023-03-07 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-03

CONDITIONS: Psychosis; Psychosocial Functioning
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental): The single treatment arm will be administered optimal health program (OHP) intervention.
  Interventions: Behavioral: Optimal Health Program

INTERVENTIONS:
Behavioral: Optimal Health Program — The OHP intervention will comprise a psychosocial management program that will be adapted to the CHR population and will be accompanied by a structured workbook. Sessions are approximately 1 hour in duration and held weekly for 6 weeks, and every two weeks for the remaining 6 weeks. The OHP has three components: 1) assessment and engagement; 2) therapy sessions, and 3) maintenance integration.

SUMMARY:
This proposal aims to adapt an evidence-based comprehensive psychosocial and mental health support program, the Optimal Health Program (OHP), to improve functioning, reduce distress, and build resiliency in youth who are at clinical risk of developing psychosis (CHR).

The main aims of the studies are 1). To adapt an existing, effective, validated psychological intervention for use in young people with CHR; 2). To evaluate the acceptability of OHP and the feasibility of conducting a clinical trial of OHP in individuals with CHR; 3). To assess the preliminary efficacy of OHP in enhancing resiliency, reducing depression and anxiety, and improving functioning in individuals with CHR in a single-arm exploratory clinical trial.

Participants will be delivered OHP intervention over 12-weeks. Measures will be completed at study entry and repeated immediately post-treatment at 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Be 16-29 years old
2. Being competent and willing to consent to study participation
3. Meets CHR criteria for a psychosis risk syndrome based on the Structured Interview for Psychosis Risk Syndromes (SIPS) either currently or at some point in the past 3 years.

Exclusion Criteria:

1. Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosis of psychotic disorder (e.g., schizophrenia spectrum disorder, mood disorder with psychotic features)
2. Diagnosis of intellectual disability previously documented in the patient chart
3. Severe developmental disorder
4. Acute suicidality requiring immediate intervention

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Adherence | post treatment (12 weeks after baseline)
  Percent sessions attended.
Retention rates | post treatment (12 weeks after baseline)
  Percent participants who complete 12-week sessions.
Attrition | post treatment (12 weeks after baseline)
  Percent participants that dropout at 12-weeks
Client Satisfaction Questionnaire | post treatment (12 weeks after baseline)
  A Likert scale from 1-4, total scores range from 8-32, with higher scores indicating greater satisfaction.

SECONDARY OUTCOMES:
Psychiatric diagnoses | baseline and post treatment (12 weeks after baseline)
  Psychiatric diagnoses will be confirmed using the Structured Clinical Interview (SCID) for DSM-5.
Connor-Davidson Resilience Scale | baseline and post treatment (12 weeks after baseline)
  This is a 25-item self-report rating scale designed to assess resilience, with higher scores indicating better outcome. Each item is rated on a 5-point scale ranging from not true at all or zero to true nearly all of the time or four. The total possible scores range from 0-100.
Structured Interview for Prodromal Symptoms | baseline and post treatment (12 weeks after baseline)
  The Structured Interview for Prodromal Symptoms (SIPS) is a widely used structured interview for diagnosing a CHR syndrome for psychosis and cases of first episode psychosis. It contains a severity rating scale (the Scale Of Psychosis-risk Symptoms, or SOPS). It is a 6-point scale, with higher scores indicating higher severity.
Calgary Depression Scale for Schizophrenia | baseline and post treatment (12 weeks after baseline)
  This scale measures the severity of depression symptoms. It is of a 4-point likert type scale with nine items with higher score indicating higher severity.
State and trait anxiety inventory | baseline and post treatment (12 weeks after baseline)
  This is a psychological inventory that measures anxiety. It consists of a 4-point likert scale with 40 items with higher scores indicating higher severity.
Global Functioning: Social | baseline and post treatment (12 weeks after baseline)
  This is a brief clinician-administered measures of social functioning, administered as a semi-structured interview with detailed anchors for ratings that address social functioning difficulties typically experienced by youth at risk for psychosis. Total possible scores on either scale ranges from 1 to 10, with higher scores indicating better social functioning.
Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) | baseline and post treatment (12 weeks after baseline)
  The MCCB includes ten tests that assess seven cognitive domains: (1) Speed of Processing; (2) Attention/Vigilance; (3) Working Memory; (4) Verbal Learning; (5) Visual Learning; (6) Reasoning and Problem Solving; and (7) Social Cognition. Requires in person administration for standardization. The test generates a raw score and a T score. Higher scores indicate better cognitive performance.
Global Functioning: Role | baseline and post treatment (12 weeks after baseline)
  This is a brief clinician-administered measures of role functioning, administered as a semi-structured interview with detailed anchors for ratings that address role functioning difficulties typically experienced by youth at risk for psychosis. Total possible scores on either scale ranges from 1 to 10, with higher scores indicating better role functioning.

OTHER OUTCOMES:
The Self-report World Health Organization - Disability Assessment Schedule (WHO-DAS 2.0) | baseline and post treatment (12 weeks after baseline)
  A 12-item generic assessment self-administered instrument for health and disability. It consists of a 5-point likert scale with higher scores indicating higher severity of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Omair Husain, MBBS, Principal Investigator — center of addiction and mental health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin A, Wood SJ, Nelson B, Beavan A, McGorry P, Yung AR. Outcomes of nontransitioned cases in a sample at ultra-high risk for psychosis. Am J Psychiatry. 2015 Mar 1;172(3):249-58. doi: 10.1176/appi.ajp.2014.13030418. Epub 2014 Nov 7. PMID 25727537
- [Background] Taylor PJ, Hutton P, Wood L. Are people at risk of psychosis also at risk of suicide and self-harm? A systematic review and meta-analysis. Psychol Med. 2015 Apr;45(5):911-26. doi: 10.1017/S0033291714002074. Epub 2014 Oct 9. PMID 25298008
- [Background] Fusar-Poli P, Nelson B, Valmaggia L, Yung AR, McGuire PK. Comorbid depressive and anxiety disorders in 509 individuals with an at-risk mental state: impact on psychopathology and transition to psychosis. Schizophr Bull. 2014 Jan;40(1):120-31. doi: 10.1093/schbul/sbs136. Epub 2012 Nov 22. PMID 23180756
- [Background] Alvarez-Jimenez M, Gleeson JF, Henry LP, Harrigan SM, Harris MG, Killackey E, Bendall S, Amminger GP, Yung AR, Herrman H, Jackson HJ, McGorry PD. Road to full recovery: longitudinal relationship between symptomatic remission and psychosocial recovery in first-episode psychosis over 7.5 years. Psychol Med. 2012 Mar;42(3):595-606. doi: 10.1017/S0033291711001504. Epub 2011 Aug 19. PMID 21854682
- [Background] McGorry PD, Hartmann JA, Spooner R, Nelson B. Beyond the "at risk mental state" concept: transitioning to transdiagnostic psychiatry. World Psychiatry. 2018 Jun;17(2):133-142. doi: 10.1002/wps.20514. PMID 29856558
- [Background] Devoe DJ, Farris MS, Townes P, Addington J. Interventions and social functioning in youth at risk of psychosis: A systematic review and meta-analysis. Early Interv Psychiatry. 2019 Apr;13(2):169-180. doi: 10.1111/eip.12689. Epub 2018 Jun 25. PMID 29938910
- [Background] Beck K, Andreou C, Studerus E, Heitz U, Ittig S, Leanza L, Riecher-Rossler A. Clinical and functional long-term outcome of patients at clinical high risk (CHR) for psychosis without transition to psychosis: A systematic review. Schizophr Res. 2019 Aug;210:39-47. doi: 10.1016/j.schres.2018.12.047. Epub 2019 Jan 14. PMID 30651204
- [Background] Gilbert MM, Chamberlain JA, White CR, Mayers PW, Pawsey B, Liew D, Musgrave M, Crawford K, Castle DJ. Controlled clinical trial of a self-management program for people with mental illness in an adult mental health service - the Optimal Health Program (OHP). Aust Health Rev. 2012 Feb;36(1):1-7. doi: 10.1071/AH11008. PMID 22513012
- [Background] Pytel' AIa, Goligorskii SD. [Treatment of chronic pyelonephritis]. Sov Med. 1972 Mar;35(3):7-13. No abstract available. Russian. PMID 5018180
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] Miller TJ, McGlashan TH, Rosen JL, Cadenhead K, Cannon T, Ventura J, McFarlane W, Perkins DO, Pearlson GD, Woods SW. Prodromal assessment with the structured interview for prodromal syndromes and the scale of prodromal symptoms: predictive validity, interrater reliability, and training to reliability. Schizophr Bull. 2003;29(4):703-15. doi: 10.1093/oxfordjournals.schbul.a007040. PMID 14989408
- [Background] Major BJ, Busuttil BE, Frauman AG. Graves' ophthalmopathy: pathogenesis and clinical implications. Aust N Z J Med. 1998 Feb;28(1):39-45. doi: 10.1111/j.1445-5994.1998.tb04457.x. No abstract available. PMID 9544385
- [Derived] Husain MO, Hawke LD, Lu Y, Kozloff N, Strudwick G, Kiang M, Wang W, Castle D, Foussias G. A mixed-methods study to evaluate the feasibility and preliminary efficacy of delivering the optimal health program (OHP) for youth at clinical high risk (CHR) for psychosis: A study protocol. PLoS One. 2024 Jul 18;19(7):e0306968. doi: 10.1371/journal.pone.0306968. eCollection 2024. PMID 39024237